CLINICAL TRIAL: NCT07343622
Title: Robot/Laparoscopic-Assisted Transanal Transection Duhamel Versus Modified Soave Pull-Through for Total Colonic Hirschsprung Disease: A Multicenter Controlled Trial
Brief Title: Robot/Laparoscopic-Assisted Transanal Transection Duhamel Versus Modified Soave Pull-Through for TCA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zunyi Medical College (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The First Affiliated Hospital of Zhengzhou University (Other); Shenzhen Longhua District Maternity and Child Healthcare Hospital (Unknown); The Affiliated Hospital of Binzhou Medical College (Unknown); Guizhou Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Zebing Zheng, Affiliated Hospital of Zunyi Medical University, Zunyi Medical College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCA/total colonic aganglionosi; No. MS-2025-406 (Other Grant/Funding Number: Guizhou provincial basic research program)
Record Dates: First submitted 2026-01-01; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Total Colonic Aganglionosis; Hirschsprung Disease; Duhamel; Soave
Keywords: Robotic surgery; total colonic aganglionosis; modified Duhamel procedure; modified Soave procedure; Hirschsprung disease
MeSH Terms: conditions — Hirschsprung Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transanal Transection Duhamel Pull-Through for total colonic aganglionosis (Experimental): Arm A: Robot-Assisted Transanal Transection Duhamel (Modified Duhamel)
  Procedure: Robot-assisted or laparoscopic-assisted abdominal mobilization (as per center standard) plus transanal external transection Duhamel pull-through with retrorectal channel creation and side-to-side colorectal/coloanal anastomosis according to a standardized operative protocol.
  Perioperative care: Standardized bowel preparation (if used), antibiotic prophylaxis, postoperative feeding pathway, and anal dilatation schedule per protocol.
  Interventions: Procedure: Transanal Transection Duhamel operation
- Modified Soave Pull-Through for total colonic aganglionosis (Active Comparator): Arm B: Modified Soave Pull-Through
  Procedure: Minimally invasive (laparoscopic or robot-assisted per center capability) mobilization plus modified Soave endorectal pull-through with mucosectomy/cuff management according to a standardized operative protocol.
  Perioperative care: Same enhanced recovery and dilatation protocol framework.
  Interventions: Procedure: Modified Soave Pull-Through

INTERVENTIONS:
Procedure: Transanal Transection Duhamel operation — The modified Duhamel procedure was performed using a transanal external rectal transection technique. Following mobilization of the ganglionated colon, the distal rectum was transected externally through the anal canal, expanding pelvic operative space and improving exposure compared with conventional pelvic transection. A retrorectal channel was created, and the colon was pulled through posterior to the native rectum. Residual rectal septum (spur) was eliminated using a transanal external compression technique, enabling a wide side-to-side colorectal or coloanal anastomosis. The anterior rectal wall was preserved, maintaining rectal sensory structures and avoiding circumferential endorectal dissection as used in Soave procedures. This approach was intended to optimize anastomotic configuration and postoperative bowel function.
  Arms: Transanal Transection Duhamel Pull-Through for total colonic aganglionosis
Procedure: Modified Soave Pull-Through — The modified Soave procedure was performed as a definitive pull-through following neonatal enterostomy. At approximately 1 year of age or older, patients underwent minimally invasive colectomy using a robotic-assisted or laparoscopic approach. The entire aganglionic colon was resected, and an endorectal pull-through was performed. The terminal ileum was delivered through the rectal cuff and anastomosed to the anal canal to restore intestinal continuity. This technique eliminates the aganglionic colorectal segment and avoids creation of a retrorectal pouch. Perioperative management and postoperative care were standardized across participating centers according to the study protocol.
  Arms: Modified Soave Pull-Through for total colonic aganglionosis

SUMMARY:
Total colonic Hirschsprung disease (TCA) is the most severe form of Hirschsprung disease and is commonly managed with neonatal enterostomy followed by delayed definitive pull-through. Despite widespread use, the optimal reconstructive procedure for TCA remains uncertain. The Duhamel and modified Soave pull-through procedures are the two most frequently adopted techniques, each with distinct theoretical advantages and limitations regarding bowel function, enterocolitis risk, and anorectal physiology. With the increasing application of minimally invasive and robot-assisted surgery, both procedures have been further refined; however, robust comparative evidence, particularly for total colonic disease, is lacking. To date, no multicenter study has provided a detailed comparison of postoperative functional outcomes and Hirschsprung-associated enterocolitis between transanal transection Duhamel and modified Soave procedures. This multicenter study compares robot-assisted transanal transection Duhamel and modified Soave pull-through in patients with pathologically confirmed TCA after neonatal enterostomy, focusing on postoperative bowel function and enterocolitis incidence.

DETAILED DESCRIPTION:
Total colonic Hirschsprung disease (TCA), also referred to as total colonic aganglionosis, represents the most severe phenotype of Hirschsprung disease and remains a major surgical challenge. Owing to extensive aganglionosis, poor nutritional status, and high risk of enterocolitis in the neonatal period, the current standard of care in most centers consists of neonatal enterostomy followed by a delayed definitive pull-through as a second-stage procedure. Despite advances in minimally invasive techniques, the optimal reconstructive strategy for TCA has not been established.

Among available options, the Duhamel procedure and the modified Soave pull-through are the two most commonly adopted techniques. The Duhamel approach, particularly when combined with a transanal external transection, preserves a retrorectal colonic reservoir, which may reduce anastomotic tension and theoretically improve postoperative bowel function. However, concerns remain regarding fecal stasis, residual spur formation, and the potential risk of postoperative enterocolitis. In contrast, the modified Soave procedure achieves complete endorectal pull-through and eliminates the aganglionic rectal segment, but it may be associated with a higher incidence of anastomotic stricture, cuff-related obstruction, and impaired anorectal motility, especially in patients with extensive disease such as TCA.

With the increasing adoption of robot-assisted and laparoscopic techniques, both procedures have been refined; nevertheless, direct comparative data evaluating functional outcomes, Hirschsprung-associated enterocolitis, and perioperative parameters between transanal transection Duhamel and modified Soave procedures-particularly in total colonic disease-remain scarce. To date, no multicenter study has provided a detailed, standardized comparison of these two surgical strategies in patients with pathologically confirmed TCA.

Therefore, this multicenter study aims to compare robot-assisted transanal transection Duhamel and modified Soave pull-through in patients with total colonic Hirschsprung disease who underwent neonatal enterostomy, with a primary focus on postoperative bowel function and the incidence of Hirschsprung-associated enterocolitis.

ELIGIBILITY:
Inclusion Criteria:

1. Definitive diagnosis of total colonic Hirschsprung disease confirmed by pathology from biopsy at neonatal enterostomy, consistent with total colonic aganglionosis.
2. Two-stage surgical strategy: neonatal enterostomy performed first, followed by definitive pull-through as a second-stage procedure.
3. Planned definitive reconstruction by one of the following techniques:
4. Robot-assisted transanal transection Duhamel, orModified Soave pull-through (minimally invasive abdominal phase allowed).
5. Availability for follow-up assessments and outcomes collection per protocol.

Exclusion Criteria:

1. Trisomy 21 (Down syndrome).
2. Definitive surgery performed by open laparotomy approach or Swenson procedure.
3. One-stage primary pull-through without neonatal enterostomy (single-stage definitive management).

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative bowel function | From enrollment to the end of treatment at 24 months
  Defecation function will be evaluated using the Rintala scoring, which comprises seven domains: bowel control, awareness of the urge to defecate, defecation frequency, stool consistency, fecal soiling, constipation, and social functioning. A total score of 17-20 points is classified as excellent, 12-16 points as good, 9-11 points as fair, and ≤8 points as poor.24 months after definitive pull-through .
Hirschsprung-associated enterocolitis (HAEC) incidence | From enrollment to the end of treatment at 24 months
  HAEC diagnosed using a standardized criterion ( prespecified clinical criteria) and recorded as:
  cumulative incidence, number of episodes, episodes requiring hospitalization/IV antibiotics.

SECONDARY OUTCOMES:
Operative time | During surgery
  During definitive pull-through operation
Intraoperative blood loss （ml） | During surgery
Postoperative length of stay (days) | From enrollment to the end of treatment at 24 months
postoperative complications | within 30 days and within 12 months
  Overall postoperative complications within 30 days and within 12 months:
  anastomotic stricture, postoperative bleeding, perianal dermatitis, other prespecified surgical complications (ileus, pelvic abscess, reoperation)
Number of anal dilatations | within 6 and 12 months
  Number of anal dilatations required (count) within 6 and 12 months
Anal resting pressure | From enrollment to the end of treatment at 24 months
  Anal resting pressure measured by anorectal manometry (mmHg) at a standardized postoperative time point (6 months, 12 months and 24 months).
Dehydration episodes | From enrollment to the end of treatment at 24 months
  Dehydration episodes (count) requiring medical intervention within 24 months.
Hospital readmissions | From enrollment to the end of treatment at 24 months
  Hospital readmissions (count) within 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Saotao Tang, M.D, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Minford JL, Ram A, Turnock RR, Lamont GL, Kenny SE, Rintala RJ, Lloyd DA, Baillie CT. Comparison of functional outcomes of Duhamel and transanal endorectal coloanal anastomosis for Hirschsprung's disease. J Pediatr Surg. 2004 Feb;39(2):161-5; discussion 161-5. doi: 10.1016/j.jpedsurg.2003.10.004. PMID 14966732
- [Background] Bhandarkar K, De Coppi P, Cross K, Blackburn S, Curry J. Long-Term Functional Outcomes and Multidisciplinary Management after Ileorectal Duhamel Pull-Through for Total Colonic Aganglionosis-20-Year Experience in a Tertiary Surgical Center. Eur J Pediatr Surg. 2024 Oct;34(5):423-429. doi: 10.1055/a-2181-2065. Epub 2023 Sep 25. PMID 37748721
- [Background] Zhang X, Cao GQ, Tang ST, Chang XP, Li S, Yang L, Li K, Zhou Y, Yang DH. Laparoscopic-assisted Duhamel procedure with ex-anal rectal transection for total colonic aganglionosis. J Pediatr Surg. 2018 Mar;53(3):531-536. doi: 10.1016/j.jpedsurg.2017.06.009. Epub 2017 Jun 27. PMID 28705638
- [Background] Halaweish I, Srinivas S, Farooqui Z, Sutthatarn P, Campbell D, Frischer J, Wood RJ, Langer JC. Duhamel Versus Swenson Pull-Through for Total Colonic Aganglionosis: A Multi-Institutional Study. J Pediatr Surg. 2024 Feb;59(2):216-219. doi: 10.1016/j.jpedsurg.2023.10.017. Epub 2023 Oct 18. PMID 37973423